CLINICAL TRIAL: NCT03997162
Title: Gastric Cancer Enhanced Recovery After Surgery Pathway
Brief Title: Early Recovery After Surgery Protocol in Improving Quality of Life in Participants With Stage 0-IIIC Gastric Cancer Undergoing Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 17482; NCI-2018-01639 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17482 (Other: City of Hope Comprehensive Cancer Center)
Record Dates: First submitted 2018-08-06; First posted 2019-06-25 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Clinical Stage 0 Gastric Cancer AJCC v8; Clinical Stage I Gastric Cancer AJCC v8; Clinical Stage II Gastric Cancer AJCC v8; Clinical Stage IIA Gastric Cancer AJCC v8; Clinical Stage IIB Gastric Cancer AJCC v8; Clinical Stage III Gastric Cancer AJCC v8; Gastric Adenocarcinoma; Pathologic Stage 0 Gastric Cancer AJCC v8; Pathologic Stage I Gastric Cancer AJCC v8; Pathologic Stage IA Gastric Cancer AJCC v8; Pathologic Stage IB Gastric Cancer AJCC v8; Pathologic Stage II Gastric Cancer AJCC v8; Pathologic Stage IIA Gastric Cancer AJCC v8; Pathologic Stage IIB Gastric Cancer AJCC v8; Pathologic Stage III Gastric Cancer AJCC v8; Pathologic Stage IIIA Gastric Cancer AJCC v8; Pathologic Stage IIIB Gastric Cancer AJCC v8; Pathologic Stage IIIC Gastric Cancer AJCC v8
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (ERAS protocol): Participants complete standard of care early recovery after surgery protocol beginning the day before surgery to day 6 after surgery.
  Interventions: Other: Best Practice; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Complete standard of care enhanced recovery after surgery protocol
  Other Names: standard of care; standard therapy
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well an early recovery after surgery protocol works in enhancing quality of life in participants with stage 0-IIIC gastric cancer undergoing surgery. The early recovery after surgery protocol may decrease pain and nausea, promote bowl function, decrease the number of days hospitalized, and improve a participant's ability to function normally after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine how the enhanced recovery after surgery (ERAS) protocol affects patient?s length of hospital stay after radical gastrectomy.

II. Determine the association between ambulation (number of steps taken) while hospitalized and complications.

III. Determine the association between pre-operatively and postoperatively drawn biochemical markers and complications, disease free survival, and overall survival.

OUTLINE:

Participants complete standard of care early recovery after surgery protocol beginning the day before surgery to day 6 after surgery.

After completion of study, participants are followed up at days 14, 30, 80-110, and 170-200, and at 11-14 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients to be included are those with a biopsy proven diagnosis of gastric adenocarcinoma who are undergoing curative gastric surgery or prophylactic total gastrectomy for genetic risk.
* Patients with clinical stage 0-IIIC will be included.
* Any performance status and any life expectancy.
* The effects of gastric surgery on the developing fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for six months following duration of study participation. Should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately.
* All subjects must have the ability to understand and the willingness to sign a written informed consent.
* Prior therapy will not be used as a limitation in this study.

Exclusion Criteria:

* Patients will be excluded if they are not candidates for surgery
* Patients will be excluded from the study if they have had prior gastric surgery, with the exception of a gastrostomy tube.
* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a biopsy proven diagnosis of gastric adenocarcinoma who are undergoing curative gastric surgery or prophylactic total gastrectomy for genetic risk
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2026-02-04 (Estimated)

PRIMARY OUTCOMES:
Length of stay | from date of surgery to discharge from hospital, assessed up to 30 days
  Will determine the length of hospital stay after surgery
Rate and type of post-operative complications | Up to 1 year

SECONDARY OUTCOMES:
Overall quality of life assessment | One time within 30 days of surgery, One time within 30 days after surgery, One time at 3 months after surgery, One time 6 months after surgery, One time 12 months after surgery
  EORTC QLQ-C30 questionnaires to measure Quality of life
QoL after stomach cancer surgery | One time within 30 days of surgery, One time within 30 days after surgery, One time at 3 months after surgery, One time 6 months after surgery, One time 12 months after surgery
  STO22 questionnaires to measure stomach cancer surgery related QoL

OTHER OUTCOMES:
Ambulation | From time of surgery to first postoperative clinic visit, assessed up to 30 days
  Number of steps taken after surgery as measured by a podometer
Immune biomarkers | one time 30 days within surgery, One time 1 day after surgery, One time 3 days after surgery, One time 30 days after surgery, One time 90 days after surgery, one time 6 months after surgery, One time 12 months after surgery
  Blood levels of hsCRP will be measured before and after surgery to determine its relationship to complications and recurrence
Disease free survival of enrolled patients | Up to 14 months after surgery
Overall survival of enrolled patients | Up to 14 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yanghee Woo, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States